CLINICAL TRIAL: NCT03984864
Title: Patient Preference Effect on Adherence and Efficacy of Exercise for Non-specific Low Back Pain
Brief Title: Preference, Exercise Therapy Adherence and Efficacy Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ariel University (Other)
Responsible Party: Principal Investigator, Shmuel Springer, Head, Physical Therapy Department, Ariel University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AU-HEA-SS-20190522
Record Dates: First submitted 2019-06-10; First posted 2019-06-13 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Low Back Pain, Recurrent
MeSH Terms: conditions — Low Back Pain | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise therapy Chosen (Experimental)
  Interventions: Other: Exercise therapy
- Exercise therapy no Chosen (Active Comparator)
  Interventions: Other: Exercise therapy

INTERVENTIONS:
Other: Exercise therapy — 3-4 items from a list of 10 general exercises - intended for treatment of low back pain

SUMMARY:
Background: Low back pain, mainly nonspecific (NSLBP) is a major cause of pain and disability worldwide. Exercise therapy (ET) is considered as the first line treatment, and it is one of the treatment modalities most commonly used by physiotherapists. Yet, ET is reliant on the adherence of patients to its various components. Research has demonstrated a positive relationship between adherence to rehabilitation programs and recovery from a variety of musculoskeletal conditions. Therefore, factors that strengthen adherence to ET may increase its efficacy for NSLBP. Converging evidence from recent studies suggest that control and choice may increase adherence to various treatments.

Therefore, the purpose of this study is to evaluate the effect of patient choice and preference on adherence and efficacy of exercise for recovery from NSLBP.

Design: Matched case control study. Participants: Fifty subjects with chronic (>3 months) NSLBP. Twenty-five participants will be allocated to exercise by preference group, and 25 aged and gender controls will be allocated to exercise group.

Inclusion criteria:

1. Non-specific low back pain (pain or discomfort in the lumbosacral area, with or without symptoms to the lower extremities), diagnosed by general physician or orthopedic surgeon.
2. Age 18-35
3. Chronic pain (greater than 3 months' duration).

Exclusion Criteria:

1. Specific cause for LBP (rheumatic diseases, tumors, fractures, fibromyalgia, previous spinal surgery, pregnancy, low back pain after car or work accidents).
2. Previous (last three years) ET treatment for NSLBP.
3. Regularly performing exercise more than WHO's recommendation:

   * 150 minutes of moderate-intensity aerobic physical activity throughout the week or at least 75 minutes of vigorous-intensity aerobic physical activity throughout the week or an equivalent combination of moderate- and vigorous-intensity activity.
   * Muscle-strengthening activities should be done involving major muscle groups on 2 or more days a week.

Procedure: After initial assessment, participants in the intervention group will be asked to choose 3-4 items from a list of 10 general exercises - intended for treatment of low back pain. Each matched participant in the control group will receive the same exercise (without the option to choose). Participants will be instructed to perform their exercises three times a week, for a period of four weeks (12 sessions total).

Outcomes: Oswestry Disability Index (ODI) Henry-Eckert Performance Assessment Tool (HEPA) Both measurements will be taken on the first and last meeting. Additionally, each participant will fill a personal weekly exercise log (selecting between complete \ incomplete \ lack of execution) - sent by e-mail.

ELIGIBILITY:
Inclusion Criteria:

1. Non-specific low back pain (pain or discomfort in the lumbosacral area, with or without symptoms to the lower extremities), diagnosed by general physician or orthopedic surgeon.
2. Age 18-35
3. Chronic pain (greater than 3 months' duration).

Exclusion Criteria:

1. Specific cause for LBP (rheumatic diseases, tumors, fractures, fibromyalgia, previous spinal surgery, pregnancy, low back pain after car or work accidents).
2. Previous (last three years) ET treatment for NSLBP.
3. Regularly performing exercise more than WHO's recommendation:

   * 150 minutes of moderate-intensity aerobic physical activity throughout the week or at least 75 minutes of vigorous-intensity aerobic physical activity throughout the week or an equivalent combination of moderate- and vigorous-intensity activity.
   * Muscle-strengthening activities should be done involving major muscle groups on 2 or more days a week.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Oswestry Disability Index (ODI) | Pre intervention/ At the end of the intervention (week four)
  Patient-completed questionnaire consisted of 10 items which gives a subjective percentage score of level of function (disability) in activities of daily living in those rehabilitating from low back pain.
  Each item consists of 6 statements scored from 0 to 5 (score of 0 indicates less disability).
  The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible
  * 0% -20%: Minimal disability
  * 21%-40%: Moderate Disability
  * 41%-60%: Severe Disability
  * 61%-80%: Crippling back pain
  * 81%-100%: These patients are either bed-bound or have an exaggeration of their symptoms Minimally clinical important difference (Johnsen et al. BMC Musculoskelet Disord. 2013) = 12.88, (sensitivity 88%, specificity 85%)

SECONDARY OUTCOMES:
Henry-Eckert Performance Assessment Tool (HEPA) | At the end of the intervention (week four)
Weekly exercise log | At the end of the intervention (week four)

CONTACTS AND LOCATIONS:
Overall Officials: shmuel springer, Principal Investigator — Ariel University; Yhonatan Levi, Study Director — Ariel University
Locations (1):
- Ariel University clininc, Ariel, Israel

IPD SHARING:
Plan to Share IPD: Undecided